CLINICAL TRIAL: NCT02093598
Title: "A Phase IIa Pharmacokinetic-pharmacodynamic Study to Confirm the Inhibitory Effect of Temsirolimus, Targeting the mTOR Pathway in Endometrial Carcinoma"
Brief Title: POEM STUDY: A Phase IIa Trial in Endometrial Carcinoma With Temsirolimus
Acronym: POEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LLO-TEM-2011-01/TEM IIG-4; 2011-005031-96 (EudraCT Number)
Record Dates: First submitted 2014-02-11; First posted 2014-03-21 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2014-03

CONDITIONS: Carcinoma, Endometrioid; mTOR Protein
Keywords: pharmacokinetic; pharmacodynamic; Carcinoma, Endometrioid; mTOR protein; temsirolimus; torisel; biological marker; phase II
MeSH Terms: conditions — Carcinoma, Endometrioid | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus (Experimental): 25 mg administered intravenously, infused over a 30- to 60-minute period once weekly for 28 days (Total doses: 4 doses).
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus
  Other Names: Torisel

SUMMARY:
Type of Application: Clinical trial of new indication.

Experimental drug: The study dose of temsirolimus will be 25 mg administered intravenously, infused over a 30- to 60-minute period once weekly for 28 days (Total doses: 4 doses). Temsirolimus is a selective inhibitor of mTOR (mammalian target of rapamycin). Pharmacotherapeutic group: Protein Kinase Inhibitors; ATC code: L01X E09.

Primary Objective:

* To identify in tumor samples future biomarkers associated with a short term exposure to temsirolimus.
* This is an exploratory clinical study. No efficacy objectives are included in this clinical trial.

Secondary Objectives:

* To estimate the tolerability for all temsirolimus-treated patients throughout the study and up to 28 days after the last dose of temsirolimus.
* To correlate observed changes with the different type of endometrial carcinoma (type I and type II), with regard to proteins related to mTOR (p4EBP1, pS6K1, c-MYC, cyclin D, p27, BAD, p53, Bcl-2 PTEN, pAKT, mTOR),
* To estimate the potential predictive value of some biomarkers (immunostaining for PTEN, pAKT, mTOR), relevant mutations in PTEN, PI3KCA, k-RAS, CTNNB1, and microsatellite instability status.
* To estimate the prognostic value of Ki67 expression after short-term presurgical therapy exposure
* To collect data about the differences in expression profile, assessed by RNA microarrays

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically-confirmed endometrial cancer
2. Stage I - II (grade 1, 2 or 3), candidates for surgery as the primary treatment
3. Age ≥ 18 years
4. WHO performance status ≤ 2
5. Adequate bone marrow function
6. Adequate liver function
7. Adequate renal function
8. Fasting serum cholesterol ≤300 mg/dL or ≤7.75 mmol/L and fasting triglycerides ≤ 2.5 x ULN
9. Signed informed consent

Exclusion Criteria:

1. Subjects who have received prior anticancer therapies for the current endometrial cancer
2. Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery or patients that may require major surgery during the course of the study
3. Prior treatment with any investigational drug within the preceding 4 weeks
4. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent
5. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
6. Uncontrolled brain or leptomeningeal metastases
7. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
8. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
9. Patients with an active, bleeding diathesis
10. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods
11. Patients who have received prior treatment with an mTOR inhibitor
12. Patients with a known hypersensitivity to rapamycine derivates or to its excipients
13. History of noncompliance to medical regimens
14. Patients unwilling to or unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the mTOR inhibitor effects of temsirolimus directly on endometrial tumor tissue after four weeks of therapy. | 1 month after last dose of the last patient
  To evaluate the mTOR inhibitor effects, assessed by level 4EBP1 and S6K1, of temsirolimus directly on endometrial tumor tissue after four weeks of therapy.

SECONDARY OUTCOMES:
To evaluate if mTOR inhibition is associated with changes in tumor-tissue | 1 month after the surgery of the last patient
  To evaluate if mTOR inhibition is associated with changes in tumor-tissue:
  * Signal transduction: AKT and PTEN
  * c-MYC, cyclin D activity
  * Proliferation index analysis: p53, p27, BAD, Bcl-2 and ki-67

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Poveda, Oncologist, Principal Investigator — Valencia, Spain
Locations (3):
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia